CLINICAL TRIAL: NCT00000355
Title: Effects of Buprenophine and Naloxone in Opiate Addicts
Brief Title: Effects of Buprenorphine and Naloxone in Opiate Addicts - 4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Pennsylvania (Other)
Purpose: Treatment
Other Study IDs: NIDA-3-0012-4; Y01-3-0012-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1995-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate the behavioral and physiological effects of buprenorphine and naloxone, both alone and in combination.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-11; Primary Completion 1996-01 (Actual); Study Completion 1996-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — PDVAMC Treatment Research Center
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States